CLINICAL TRIAL: NCT06167044
Title: Effect of Thoracic Spine Mobilization on Pain, Functional Disability and Proprioception in Patients With Lumbosacral Radiculopathy.
Brief Title: Effect of Thoracic Mobilization on Lumbar Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, aya abd elmohsen salah eldeen, aya abd elmohsen salah eldeen, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: thoracic mobilization in LR
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Lumbosacral Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thoracic mobilization group (Active Comparator): which will include 17 patients who will receive thoracic manual mobilization exercises in addition to selected physical therapy .The treatment will conducted for 45 minutes, 3 sessions per week for 6 weeks.
  Interventions: Other: thoracic mobilization
- control group (No Intervention): which will include 17 patients who will receive selected physical therapy.The treatment will conducted for 45 minutes, 3 sessions per week for 6 weeks.

INTERVENTIONS:
Other: thoracic mobilization — Thoracic mobilization will be performed for the thoracic spine mobilization group, thoracic mobilization therapy will be performed for five minutes.
  Arms: thoracic mobilization group

SUMMARY:
The purpose of the study will be to:

* To investigate the effect of thoracic mobilization on back and leg pain in patients with lumbosacral radiculopathy.
* To investigate the effect of thoracic mobilization on functional disability in patients with lumbosacral radiculopathy.
* To investigate the effect of thoracic mobilization on proprioception in patients with lumbosacral radiculopathy.

DETAILED DESCRIPTION:
To investigate the effect of thoracic mobilization on back and leg pain, functional disability and proprioception in patients with lumbosacral radiculopathy.

1-Thirty four patients of both sexes with unilateral chronic lumbar radiculopathy at L4-L5 or/ and L5-S1 levels will participate in this study. The patients will be diagnosed as having lumbar radiculopathy based on careful clinical examination by neurologist . The diagnosis will be confirmed by CT scan or MRI.

Patients will be recruited from the outpatient clinic of Faculty of Physical Therapy, Cairo University and private clinics. Patients in this study will be randomly divided into two groups.

* Group (I) which will include 17 patients who will receive manual mobilization exercises in addition to selected physical therapy .
* Group (II) which will include 17 patients who will receive selected physical therapy.

The treatment will conducted 3 sessions per week for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral chronic lumbosacral radiculopathy at L4- L5 or / and L5-S1 levels confirmed by MRI.
2. The age of patients will be ranged from 30 to 45 years.
3. Duration of pain will be more than 12 weeks.
4. Patients with a positive straight leg raising (SLR) test.
5. Patients with sufficient cognitive abilities that enables them to understand and follow instructions .
6. Patients had to report an average pain level of more than five on the Visual Analogue Scale (VAS) and a lumbar spine range of motion (ROM) of at least 50% of the accepted normal range.
7. Patients with body mass index< 30kg/m2

Exclusion Criteria:

1. Cauda equina syndrome.
2. Ankylosing spondylitis, thoracic deformities (pectus carinatum, excavatum), spina bifida, fractures, postoperative spinal conditions, diabetes, inflammatory processes.
3. Previous inner ear infection or vestibular disorder with unresolved balance disturbance, history of head trauma with residual neurological deficits.
4. Spinal tumor.
5. Previous lumbar surgery.
6. Sever musculoskeletal disease.
7. Peripheral mononeuropathies or polyneuropathy.
8. Obesity .
9. Pregnancy.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
functional disability | baseline
  we will use Oswestry Disability Index (ODI)
pain level | baseline
  we will use Visual analogue scale (VAS)
lumbar proprioception | baseline
  we will use The Biodex System 3 pro isokinetic dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Ibrahim Rehab, Assistant Professor, Study Chair — physical therapy for neuromuscular disorder and its surgery; Ebtesam Mohamed Fahmy, Professor, Study Chair — faculty of medicine; HOSSAM MOHAMMED MOHAMMED, Lecturer, Study Chair — physical therapy for neuromuscular disorder and its surgery
Locations (1):
- Faculty of Physical Therapy Cairo University, Cairo, Egypt